CLINICAL TRIAL: NCT06182072
Title: A Phase I/Ib Trial of ProAgio, an Anti- αvβ3 Integrin Cytotoxin, in Combination With Gemcitabine and Nab-paclitaxel or Gemcitabine, Nab-paclitaxel and Atezolizumab for Advanced Pancreatic Cancer
Brief Title: ProAgio in Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ProDa BioTech, LLC (Industry)
Collaborators: University of Alabama at Birmingham (Other); Georgia State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UAB 2335 v2.1
Record Dates: First submitted 2023-11-21; First posted 2023-12-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
MeSH Terms: interventions — Gemcitabine; Taxes

STUDY DESIGN:
Intervention Model Description: This study includes a dose escalation arm, followed by an expansion arm at the ideal dose for participants with previously untreated advanced Pancreatic ductal adenocarcinoma (PDAC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): ProAgio Dose Levels (DL) 1,2,3,4
  ProAgio combined with gemcitabine, and nab paclitaxel is administered to study participants by intravenous injections on days 1, 8, 15, 21 every 4-week Cycle, gemcitabine and nab paclitaxel on day 1, 8, 15 every 4-week cycle during the study.
  Other Names:
  ACT50, G-nP: Gemcitabine, nab-Paclitaxel
  Interventions: Drug: ProAgio Dose Levels (DL) 1,2,3,4; Drug: Gemcitabine, nab paclitaxel
- Standard Arm (Experimental): In cycle 1 of dose expansion phase of the study, half of patients (n=6) will be administered ProAgio only on day 1, 8, 15, 22 every 4-week Cycle, and half of patients (n=6) will be administered gemcitabine and nab paclitaxel are administered day 1, 8, 15 every 4-week cycle. In the atezolizumab containing cohort atezolizumab will be administered day 1 of cycle 1, and then will be repeated every 3 weeks.
  Other Names:
  ACT50, G-nP: Gemcitabine and nab-Paclitaxel, atezolizumab
  Interventions: Drug: ProAgio Dose Levels (DL) 1,2,3,4; Drug: Gemcitabine, nab paclitaxel

INTERVENTIONS:
Drug: ProAgio Dose Levels (DL) 1,2,3,4 — ProAgio combined with gemcitabine and nab paclitaxel (G-nP) in previously untreated subjects with metastatic PDAC.
  Other Names: ACT50
Drug: Gemcitabine, nab paclitaxel — ProAgio combined with gemcitabine and nab paclitaxel (G-nP) in previously untreated subjects with metastatic PDAC.
  Other Names: (G-nP)

SUMMARY:
This is an open-label Phase I/Ib dose-escalation, dose-expansion clinical trial of the safety, pharmacokinetics and clinical activity of ProAgio combined with gemcitabine, nab-paclitaxel (G-nP) or gemcitabine, nab-paclitaxel (G-nP) and atezolizumab in previously untreated subjects with metastatic pancreatic ductal adenocarcinoma (PDAC)

DETAILED DESCRIPTION:
This is an open-label Phase I/Ib dose-escalation, dose-expansion clinical trial of the safety, pharmacokinetics and clinical activity of ProAgio combined with gemcitabine, nab-paclitaxel (G-nP) or gemcitabine, nab-paclitaxel (G-nP) and atezolizumab in previously untreated subjects with metastatic PDAC. The study will use an EWOC design in Phase I to determine the recommended RP2D of ProAgio with gemcitabine, nab paclitaxel (G-nP) and atezolizumab. After the estimation of RP2D of ProAgio alone, the trial will continue to estimate the RP2D of ProAgio when combined with G-nP, starting from 2 dose levels lower than the estimated RP2D of ProAgio alone. EWOC design will enroll 2 subjects per cohort with 4 combination dose levels.

Subjects will be selected based on following criteria: previously untreated advanced PDAC, ECOG performance status (0-1), and adequate organ functions. Subjects with recent surgeries, history of recent thromboembolic events or significant cardiovascular disease will be excluded.

Once the MTD and RP2D of ProAgio with G-nP RP2D have been identified, an expansion cohort of 12 subjects with metastatic PDAC (n=6 receiving ProAgio and n=6 receiving ProAgio + GnP) will begin. The purpose of the expansion cohort is to confirm the safety of the regimen and provide preliminary data on the activity of both ProAgio monotherapy and ProAgio + GnP. An additional expansion cohort with ProAgio, GnP and atezolizumab will enroll patients with metastatic PDAC (n=18 including 6 patients safety run-in). The purpose of the expansion cohort is to confirm the safety of the regimen and provide preliminary data on the activity of and ProAgio, GnP and atezolizumab combination.

Data regarding adverse events will be collected, attributed and graded according to NCI CTCAE version 5.0 criteria. Pharmacokinetic and pharmacodynamic data will be collected per the study flow chart. Response will be evaluated every 2 months using RECIST criteria. Planned secondary analyses will include ORR, duration of response, PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age on day of signing informed consent.
2. Histologic or cytologic diagnosis of pancreatic adenocarcinoma with clinical stage IV.
3. In the dose escalation phase: patients must be eligible for gemcitabine and nab paclitaxel. For dose expansion phase: patients must have received 5FU-based therapy for metastatic disease or for neoadjuvant/adjuvant therapy in prior 12 months.
4. Presence of a lesion that can be safely biopsied for correlative assays.
5. Patient must meet the following laboratory values at the screening visit:

   * Absolute Neutrophil Count ≥1.5 x 10'9/L
   * Platelets ≥100 x 10'9/L
   * Hemoglobin (Hgb) ≥9 g/dL
   * Serum creatinine <1.5 mg/dL OR Creatinine Clearance ≥60 mL/min using Cockcroft-Gault formula
   * Total bilirubin ≤1.5 x ULN
   * Aspartate transaminase (AST) ≤2.5 x ULN, except for subjects with liver metastasis, who may only be included if AST ≤5.0 x ULN
   * Alanine transaminase (ALT) ≤2.5 x ULN, except for subjects with liver metastasis, who may only be included if ALT ≤5.0 x ULN
6. Presence of measurable disease by RECIST 1.1 criteria
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Written informed consent must be obtained prior to any screening procedures.
9. Normal ECG defined as the following: QTcF at screening <450 ms (male subjects), <460 ms (female subjects)
10. Before enrollment, a woman must be either:

    1. Not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 IU/mL); permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy.
    2. Of childbearing potential and practicing (during the study and for 6 months after receiving the last dose of study agent) a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: eg, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods; true abstinence (when this is in line with the preferred and usual lifestyle of the subject).
    3. Note: If the childbearing potential changes after start of the study (eg, woman who is not heterosexually active becomes active) a woman must begin a highly effective method of birth control, as described above.
11. A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at screening.
12. During the study and for 6 months after receiving the last dose of study agent, a woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction.
13. A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug.
14. Sign an informed consent document indicating that they understand the purpose of and procedures required for the study, are willing to participate in the study, and are willing and able to adhere to the prohibitions and restrictions specified in this protocol. Informed consent must be obtained before performing any study specific procedures.

Exclusion Criteria:

1. Prior exposure to gemcitabine and nab paclitaxel
2. Clinically significant peripheral neuropathy
3. Any untreated central nervous system (CNS) lesion. However, subjects are eligible if:

   a) all known CNS lesions have been treated with radiotherapy or surgery and b) patient remained without evidence of CNS disease progression ≥4 weeks after treatment.
4. Use of hematopoietic colony-stimulating growth factors (eg, G-CSF, GMCSF, M-CSF), thrombopoietin mimetics or erythroid stimulating agents ≤ 2 weeks prior start of study treatment. If erythroid stimulating agents were initiated more than 2 weeks prior to the first dose of study treatment and the patient is on a stable dose, they can be maintained.
5. Active unstable autoimmune disease. Documented history of autoimmune disease that is well controlled on stable immune suppressive therapy can be enrolled after discussion with principal investigator.
6. Allogenic bone marrow or solid organ transplant.
7. Known history or current interstitial lung disease or non-infectious pneumonitis.
8. Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers and any completely resected carcinoma in situ.
9. Clinically significant infection, including known HIV or hepatitis C infection, or known hepatitis B surface antigen positivity. Testing of asymptomatic patients will not be required.
10. Clinically significant ongoing infection.
11. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 14 days or 5 half-lives before enrollment or is currently enrolled in the treatment stage of an investigational study.
12. A woman who is pregnant or breast-feeding, or a woman who is planning to become pregnant or a man who plans to father a child while enrolled in this study or within 30 days after the last dose of study agent.
13. Had hospitalization for infection or major surgery (eg, requiring general anesthesia) within 2 weeks before enrollment or have not fully recovered from surgery. Note: subjects with surgical procedures conducted under local anesthesia may participate.
14. History or current diagnosis of cardiac disease indicating significant risk of safety for subjects participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

    1. recent myocardial infarction (within last 6 months),
    2. uncontrolled congestive heart failure,
    3. unstable angina (within last 6 months),
    4. clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker).

    Following additional exclusion criteria applies only to the patients in the cohort including atezolizumab:
15. Active or prior documented autoimmune or inflammatory disorders (including, but not limited to inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
    * Patients with type I diabetes mellitus who are on an insulin regimen are eligible for the study
16. Current or prior use of immunosuppressive medication ≤ 14 days prior to registration.

    The following are exceptions to this criterion:
    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine ≤30 days prior to registration. Note: Patients, if enrolled, should not receive live vaccine whilst on study treatment and up to 30 days after the last dose of study treatment.
18. History of pneumonitis/interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of ProAgio combined with gemcitabine and nab paclitaxel. | 2 Years
  Physical examination, vital signs, clinical laboratory evaluations (CBC, serum chemistry, coagulation studies, LFTs, and assessment of subject reported AEs (via CTCAE v5.0) and SAEs will be used to evaluate safety.
Determine the patient's height. | 2 Years
  Height measured in Centimeters (cm)
Determine the patient's weight. | 2 Years
  Weight measured in Kilograms (kg)
Determine the patient's body temperature. | 2 Years
  Body Temperature measured in Celsius
Determine the patient's Respiration Rate. | 2 Years
  Respiration Rate measured in times/min
Determine the patient's Heart Rate. | 2 Years
  Heart Rate measured in beats/min
Determine the patient's Systolic Blood Pressure | 2 Years
  Systolic Blood Pressure measured in mmHg
Determine the patient's Diastolic Blood Pressure. | 2 Years
  Diastolic Blood Pressure measured in mmHg
Determine the patient's Pulse Oximetry. | 2 Years
  Perform Pulse Oximetry measured in (SpO2)
Determine a single ideal dose which will be selected for further investigation in the dose escalation cohort. | 2 Years
  Following completion of the dose escalation cohort, all available data relating to the pharmacokinetics, pharmacodynamics, efficacy and safety of ProAgio combined with gemcitabine and nab paclitaxel will be reviewed by the study team including the Principle Investigator, clinical pharmacology collaborators and the sponsor. A single ideal dose will then be selected for further investigation in the dose escalation cohort. This ideal dose may or may not be the same as the MTD.

SECONDARY OUTCOMES:
Determine the total integrated area under the plasma drug concentration-time curve (AUC). | 2 Years
  Analyze pharmacokinetics to determine the total integrated area under the plasma drug concentration-time curve (AUC).
Determine the Peak Plasma Concentration (Cmax). | 2 Years
  Pharmacokinetics will be analyzed by determining Peak Plasma Concentration (Cmax).
Determine how well the patient eliminates the study drug (CL). | 2 Years
  Pharmacokinetics will be analyzed by determining how well the patient eliminates the drug (CL).
Determine Volume of distribution (Vd). | 2 Years
  Pharmacokinetics will be analyzed by determining Volume of distribution (Vd).
Determine the study drug half-life (t1/2). | 2 Years
  Pharmacokinetics will be analyzed by determining the study drug half-life (t1/2).
An attempt will be made to determine dose proportionality of ProAgio. | 2 Years
  Pharmacokinetics will be analyzed by determining the amount of drug reaching the systemic circulation.
Evaluate Objective response rate (ORR). | 2 Years
  Objective response rate (ORR), defined as complete response (CR) or partial response (PR) through cycle 6 per RECIST 1.1 as a proportion of n=6 of the Phase1b cohorts.
Evaluate Duration of response (DOR). | 2 Years
  Duration of response (DOR), determined from date of best response to progression or death.
Evaluate Progression-free Survival (PFS). | 2 Years
  Progression-free Survival (PFS), determined from date of 1st dose of study drug to progression or death.
Evaluate Overall Survival (OS). | 2 Years
  Overall Survival (OS) determined from date of 1st dose of study drug to death from any cause. CA19-9 will be assessed by descriptive statistics.
Evaluate patient tumor response. | 2 Years
  MR imaging assessment of patient tumor response using a unique MRI photon to monitor tumor changes and tumor blood perfusion changes.

OTHER OUTCOMES:
Evaluate patient Pyruvate kinase-M2 (PKM2). | 2 Years
  Descriptive statistics will be used to summarize the expression of PKM2 in each batch of blood samples collected from subjects at pre-treatment, 48 hrs, and 14 days post-treatment, respectively.
Evaluate tumor biology changes due to treatment. | 2 Years
  Descriptive statistics will be used to summarize the desmoplastic stroma, intratumoral collagen, blood vessels, CAPSC, and αvβ3 expression in each batch of biopsy samples taken from subjects at pre-treatment and 4 weeks post-treatment, respectively.
Evaluate patient tumor fibrosis pre and post treatment with ProAgio. | 2 Years
  Perfusion MRI will be performed pre and on treatment with ProAgio to assess impact on fibrosis.
Evaluate patient monitor tumor angiogenesis pre and post treatment with ProAgio. | 2 Years
  Perfusion MRI will be performed pre and on treatment with ProAgio to assess impact on angiogenesis.
Evaluate patient tumor blood perfusion pre and post treatment with ProAgio. | 2 Years
  Perfusion MRI will be performed pre and on treatment with ProAgio to assess impact on perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akce, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- O'Neal Comprehensive Cancer Center, University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Bandi DSR, Sarvesh S, Nagaraju GP, Kim H, Foote J, Bae S, Yoon KJ, Malla M, Masood A, Akce M, Liu ZR, El-Rayes BF. ProAgio, a Novel Integrin alphavbeta3 Targeted Cytotoxin, Suppresses Tumor Growth and Reprograms the PDAC Microenvironment. bioRxiv [Preprint]. 2026 Jan 16:2026.01.15.699725. doi: 10.64898/2026.01.15.699725. PMID 41648362